CLINICAL TRIAL: NCT00318578
Title: Prognosis Factors Associated With Convulsive Status Epilepticus in Adults: A Multicenter Cohort Study
Brief Title: Prognosis Factors Associated With Convulsive Status Epilepticus in Adults
Status: Completed | Type: Observational
Sponsor: Versailles Hospital (Other)
Other Study IDs: LEGRIEL stephane
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-08

CONDITIONS: Status Epilepticus
Keywords: convulsive status epilepticus; outcome; prognosis factors; seizure duration; adult; electroencephalogram; intensive care unit
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The aim of the study is to evaluate, prospectively, prognosis factors associated with convulsive status epilepticus (CSE) in adults hospitalized in intensive care units.

DETAILED DESCRIPTION:
Status epilepticus is a neurologic and medical emergency associated with high mortality and morbidity rates. According to the operational definition Convulsive Status Epilepticus (CSE) is defined as a single clinical seizure lasting more than 10 min, or two or more repeated seizures over a period of more than 10 minutes without intervening recovery of consciousness.

There are a few to date in literature reporting prognosis factors associated with this condition and, at this time, there are no published data considering an operational definition of CSE.

In a retrospective study considering an operational definition we identified a seizure duration of 15 min associated with poor outcome (not yet published).

The principal goal of this study is to evaluate factors associated with outcome in CSE, in particular seizure duration of more than 15 minutes.

The secondary goals are to evaluate the epidemiology and management at every stage of CSE thus redefined.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Convulsive status epilepticus according to operational definition as any seizure lasting for 10 minutes or longer, or two or more intermittent seizures lasting for greater than 10 minutes from which the patient did not regain consciousness.
* Beginning of seizure less than 12 hours before intensive care unit admission
* Convulsive status epilepticus occurring during intensive care unit stay

Exclusion Criteria:

* Less than 18 years old
* Patients that seized up to 9 minutes
* Beginning of seizure more than 12 hours before intensive care unit admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-03; Study Completion 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Stephane LEGRIEL, MD, Principal Investigator — Versailles Hospital; Bruno MOURVILLIER, MD, Principal Investigator — Centre Hospitalier Bichat Claude Bernard
Locations (34):
- France (34):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Centre Hospitalier d'Annonay, Annonay
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Robert Ballanger, Aulnay-sous-Bois
  - Centre Hospitalier Rene Dubos, Cergy-Pontoise
  - Centre Hospitalier de Chartres, Chartres
  - Centre Hospitalier de Châlons-en-Champagne, Châlons-en-Champagne
  - Centre Hospitalier Universitaire Antoine Beclere, Clamart
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier de Compiegne, Compiègne
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Centre Hospitalier de Dourdan, Dourdan
  - Centre Hospitalier de Dreux, Dreux
  - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Centre Hospitalier de Versailles, Le Chesnay
  - Centre Hospitalier Universitaire La Timone, Marseille
  - Centre Hospitalier Sambre Avesnois, Maubeuge
  - Centre Hospitalier de Meaux, Meaux
  - Centre Hospitalier Universitaire de Nancy, Nancy
  - Centre Hospitalier Pierre Bérégovoy, Nevers
  - Centre Hôspitalier ARCHET, Nice
  - Centre Hospitalier Georges Renon, Niort
  - Centre Hospitalier Universitaire d'Orléans, Orléans
  - Centre Hospitalier Universitaire Cochin, Paris
  - Centre Hospitalier Universitaire Lariboisiere, Paris
  - Centre Hospitalier Bichat Claude Bernard, Paris
  - Fondation Hopital Saint Joseph, Paris
  - Centre Hospitalier Francois Mitterrand, Pau
  - Clinique Mutualiste de Pessas, Pessac
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier de Roanne, Roanne
  - Centre Hospitalier de Rodez, Rodez
  - Centre Hospitalier Mémorail France Etats Unis Saint Lo, Saint-Lô
  - Centre Hospitalier Foch, Suresnes